CLINICAL TRIAL: NCT05210452
Title: Treatment of Alopecia Using Follicular Stem Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_FollCells
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with alopecia receiving standard treatment and follicular stem cells (Experimental): Patients with alopecia receiving standard treatment and autologous follicular stem cells
  Interventions: Biological: Follicular stem cells; Other: Standard treatment according to the clinical protocols
- Patients with alopecia receiving standard treatment (Active Comparator): Patients with alopecia receiving standard treatment
  Interventions: Other: Standard treatment according to the clinical protocols

INTERVENTIONS:
Biological: Follicular stem cells — Cultured autologous follicular stem cells
  Arms: Patients with alopecia receiving standard treatment and follicular stem cells
Other: Standard treatment according to the clinical protocols — Standard treatment of alopecia according to the clinical protocols

SUMMARY:
Treatment of alopecia using the injections of cultured stem cells from human hair follicles,(which contain epithelial and mesenchymal cells stem cell)

DETAILED DESCRIPTION:
The aim of the project is to develop a biomedical cell product based on and stem progenitor cells of the hair follicle and dermal papilla, to study its efficacy in the treatment of alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of alopecia areata, androgenic alopecia and other non-scarring hair loss
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* Acute or chronic diseases in the stage of decompensation
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding, or fertile patients who are not using adequate contraceptive methods
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of cured patients | 6 month
  Number of cured patients with significant clinical improvement
Number of cured patients | 1 year
  Number of cured patients with significant clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Zinaida Kvacheva, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus

IPD SHARING:
Plan to Share IPD: No